CLINICAL TRIAL: NCT04887623
Title: Dynamics of Nucleocapsid Antigen Serum Levels and Other Markers of Infection and Inflammation in Hospitalized Coronavirus Disease 2019 (COVID-19) Patients - a Pilot Study
Brief Title: Dynamics of Markers of Infection and Inflammation in Hospitalized Coronavirus Disease 2019 (COVID-19) Patients
Status: Recruiting | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, principal investigator, University Hospital Hradec Kralove
Other Study IDs: UHHK042021
Record Dates: First submitted 2021-03-27; First posted 2021-05-14 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Covid19; Interleukin 6; viremia; nucleocapsid antigen
MeSH Terms: conditions — COVID-19; Viremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients requiring admission to the hospital due to a moderate and severe COVID-19 infection may differ in their ability to respond to viral infection and to eliminate viral load.

Several comorbidities and interventions like antivirotic or antiinflammatory treatment may also modify expected patients response and decrease of viral load.

In this observational study, evolution of selected inflammatory markers, indicators of severity of infection and patient characteristics will be followed and recorded in hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
In this pilot study, 30 consecutive COVID-19 patients requiring admission to the hospital due to a moderate and severe COVID-19 infection will be included into an observational study.

Following parameters will be recorded: age, sex, weight, height, comorbidities, smoking habit,spiritus and drug intake history, length of COVID-19 symptoms, clinical and laboratory parameters, the use of different COVID-19 intervention (remdesivir, convalescent plasma, monoclonal antibodies, corticosteroids, tocilizumab and other medication), used initial and maximal organ support during the stay and outcome of the stay in the hospital and 28th and 90th day, laboratory markers of severity of infection - serum and tracheal aspirate (in ventilated patients) levels of nucleocapsid antigen,Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV2) viremia and quantity in tracheal aspirates (in ventilated patients), makers of inflammatory response (C- reactive proteins, Interleukin 6, procalcitonin, ferritin) and selected other biochemical values (blood count, D-dimers, flow cytometry).

ELIGIBILITY:
Inclusion Criteria:

* SARS CoV2 positive test within last 14 day
* bilateral infiltrates on chest X.ray or CT
* need for oxygen to keep pulse oximetry saturation above 92% or other respiratory support measures (HFNO, non-invasive ventilation or invasive ventilation)

Exclusion Criteria:

* known history of intersticial lung disease
* known history of congestive heart failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized COVID-19 with moderate to severe course of COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prediction of severity of lung dysfunction based on initial nucleocapsid antigen serum levels | Admission
  Correlation between baseline nucleocapsid serum levels and the Ordinal Scale for Clinical Improvement
Prediction of severity of lung dysfunction based on initial interleukin-6 serum levels | Admission
  Correlation between baseline interleukin -6 serum levels and Ordinal Scale for Clinical Improvement
Prediction of severity of lung dysfunction based on | Admission
  Correlation between baseline CRP serum levels and Ordinal Scale for Clinical Improvement

SECONDARY OUTCOMES:
Effect of the dose of corticosteroids on the nucleocapsid antigen serum levels | up to 28 days
  Correlation between the dose of corticosteroids and evolution of nucleocapsid serum levels
Effect of the remdesivir on the nucleocapsid antigen serum levels | up to 28 days
  Comparison of the nucleocapsid antigen serum levels between patients receiving and not receiving remdesivir
Effect of comorbidities on persistence of tracheal viral load assessed using tracheal aspirate semiquantitative PCR | up to 28 days
  Analysis of the effect of comorbidities on evolution of viral load assessed using tracheal aspirate semiquantitative PCR
Effect of age on persistence of tracheal viral load assessed using tracheal aspirate semiquantitative PCR | up to 28 days
  Analysis of the effect of age on evolution of viral load assessed using tracheal aspirate semiquantitative PCR
Effect of age on viral load assesed using nucleocapsid antigen serum levels | up to 28 days
  Analysis of the effect of age on evolution of nucleocapsid antigen serum levels
Effect of comorbidities on viral load assessed using nucleocapsid antigen serum levels | up to 28 days
  Analysis of the effect of comorbidites on evolution of nucleocapsid antigen serum levels
Tracheal viral load quantification using tracheal nucleocapsid antigen | up to 28 days
  Correlation between the number of cycles of amplification of real time PCR and nucleocapsid antigen tracheal aspirate levels and between the number of cycles of amplification of real time PCR and nucleocapsid antigen serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Palicka, MD, CSc., Study Chair — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Undecided